CLINICAL TRIAL: NCT00751764
Title: An Open-Label, Single-Dose Study to Evaluate the Excretion of Moxidectin Into the Breast Milk of Lactating, Non-breastfeeding Women.
Brief Title: Study Evaluating The Excretion Of Moxidectin Into The Breast Milk Of Lactating, Non-Breastfeeding Women
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Wyeth (Registry Contact: Clinical Trial Registry Specialist), Wyeth
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: 3110A1-1002
Record Dates: First submitted 2008-09-11; First posted 2008-09-12 (Estimated); Last update posted 2010-09-16 (Estimated); Status verified 2010-09

CONDITIONS: Infection
MeSH Terms: conditions — Infections | interventions — moxidectin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Moxidectin

INTERVENTIONS:
Drug: Moxidectin

SUMMARY:
The purpose of this study is to evaluate the extent of moxidectin transfer into the breast milk of lactating women and to provide the initial pharmacokinetic and safety profile of moxidectin in lactating women.

ELIGIBILITY:
Inclusion criteria:

Healthy lactating women aged 21 to 45 years inclusive at screening. Women should:

* Be at least 12-weeks postpartum after uncomplicated delivery with a full milk supply established.
* Be willing to discontinue breastfeeding permanently and should be in the process of weaning their infant. Care should be taken to ensure that subjects have not discontinued breastfeeding an infant in order to participate in the study.
* Not plan to breastfeed within 9 months of study drug administration.
* Be willing to fully express breast milk from both breasts during the duration of the milk collection portion of the study. Subjects must be able to express milk from each breast at each pumping session using a breast pump.
* Body mass index in the range of 18 to 35 kg/m2.

Exclusion criteria:

* Presence or history of any disorder that may prevent the successful completion of the study.
* Any significant cardiovascular, hepatic, renal, respiratory, gastrointestinal, endocrine, immunologic, dermatologic, hematologic, neurologic, or psychiatric disease.

Ages: 21 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2008-11; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Blood samples | 4 months

SECONDARY OUTCOMES:
Safety based on adverse event monitoring, vital sign measurements, 12-lead ECGs and routine lab tests. | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (1):
- Plymouth, United Kingdom